CLINICAL TRIAL: NCT04827602
Title: Drug Allergy Labels in Different Electronic Health Records After Drug Allergy Investigation
Brief Title: Drug Allergy Labels After Drug Allergy Investigation
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Research Unit Of General Practice, Copenhagen (Other)
Responsible Party: Principal Investigator, Sara Fransson, Ph.D student, University Hospital, Gentofte, Copenhagen
Other Study IDs: GEH-R-20068776
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Drug Hypersensitivity
Keywords: drug allergy; drug allergy labels; penicillin allergy labels
MeSH Terms: conditions — Drug Hypersensitivity | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergy tested group: Patients who have completed penicillin allergy testing
  Interventions: Other: Drug allergy label status in electronic health records

INTERVENTIONS:
Other: Drug allergy label status in electronic health records — Registered drug allergy labels in primary care and hospital electronic medical charts

SUMMARY:
The aim of this study is to investigate the degree of match between the drug allergy label in the hospital's electronic health record and primary care's electronic health record among patients who previously have been drug allergy tested.

DETAILED DESCRIPTION:
Patients who previously have been penicillin allergy tested in 2017 to 2019 at the Allergy Clinic at Gentofte Hospital is included in the study. Patients are identified through a drug allergy database at the department.

A letter describing the study and the data collection process will be sent to the patients' General Practice offices (GP).

Data collection: The patients GP's are contacted by telephone where the information about the drug allergy labels in their electronical medical charts are shared. On the same day as the phone contact to the GP's office, the patient's electronical health record in the hospital system is accessed in order to gain information about the current drug allergy registrations.

Predictors for the explanatory analysis is collected partly through the phone call to the GP (such as numbers of patients and physicians at each GP and the electronic health system used), from the hospital electronic health record (such as number of hospital admissions since drug allergy testing) and from the drug allergy database.

ELIGIBILITY:
Inclusion Criteria:

* Penicillin allergy tested at the Allergy Clinic, Copenhagen University Hospital - Herlev and Gentofte, Copenhagen, Denmark in 2017-2019

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients who completed penicillin allergy testing in 2017 to 2019 at the Allergy Clinic, Copenhagen University Hospital - Herlev and Gentofte, Copenhagen, Denmark. The study population is estimated to 900 participants from both the Capital Region and Region Zealand.
Sampling Method: Non-Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Degree of matching drug allergy testing and drug allergy labels | Baseline
  Degree of match between allergy testing outcomes and registered drug allergy labels in primary care and hospital electronic health records

SECONDARY OUTCOMES:
Degree of match between registered drug allergy labels | Baseline
  Degree of match between registered drug allergy labels in primary care and hospital electronic health records

OTHER OUTCOMES:
Analysis of predictors for failure to update drug allergy labels | Baseline
  Exploratory analysis of predictors for failure to update the drug allergy labels. Predictors include sex, age, immediate/delayed index allergic reaction, drug allergy test results, patients pr GP, doctors pr GP, electronic system used, drug allergy test referrals from the same GP, drug allergy labels pr patient and admissions since drug allergy testing pr patient.

CONTACTS AND LOCATIONS:
Overall Officials: Lene H. Garvey, Principal Investigator — Allergy Clinic, Copenhagen University Hospital, Copenhagen
Locations (1):
- Allergy Clinic, Department of Dermato-Allergology, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lachover-Roth I, Sharon S, Rosman Y, Meir-Shafrir K, Confino-Cohen R. Long-Term Follow-Up After Penicillin Allergy Delabeling in Ambulatory Patients. J Allergy Clin Immunol Pract. 2019 Jan;7(1):231-235.e1. doi: 10.1016/j.jaip.2018.04.042. Epub 2018 May 22. PMID 29800754
- [Result] Vyles D, Chiu A, Routes J, Castells M, Phillips EJ, Kibicho J, Brousseau DC. Antibiotic Use After Removal of Penicillin Allergy Label. Pediatrics. 2018 May;141(5):e20173466. doi: 10.1542/peds.2017-3466. PMID 29678929
- [Result] Sacco KA, Bates A, Brigham TJ, Imam JS, Burton MC. Clinical outcomes following inpatient penicillin allergy testing: A systematic review and meta-analysis. Allergy. 2017 Sep;72(9):1288-1296. doi: 10.1111/all.13168. Epub 2017 Apr 26. PMID 28370003